CLINICAL TRIAL: NCT02925208
Title: Radiological Classification of the Vertical Segment of Facial Nerve in Cochlear Implant Surgery
Brief Title: Radiological Classification of the Facial Nerve
Status: Completed | Type: Observational
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Other Study IDs: ENT_1_10_2016
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Severe to Profound Sensorineural Hearing Loss; Undergoing Cochlear Implant Surgery

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cochlear Implant: Patients with severe to profound sensorineural hearing loss who underwent cochlear implant surgery
  Interventions: Other: cochlear implant surgery

INTERVENTIONS:
Other: cochlear implant surgery — patients with severe to profound sensorineural hearing loss who underwent cochlear implant surgery

SUMMARY:
Cortical mastoidectomy and posterior tympanotomy is a classic approach for cochlear implant. Intimate knowledge of the relevant surgical anatomy of the temporal bone and facial recess is important to safely perform the posterior tympanotomy. Anatomical variation of facial nerve such as lateral or anterior position of vertical segment of facial nerve, will render this approach challenging. In this research, investigators proposed a Radiological Classification system of the position of vertical segment of facial nerve in relation to the lateral semicircular canal to predict difficult cases with narrow facial recess.

DETAILED DESCRIPTION:
Cochlear implantation done by mastoidectomy, posterior tympanotomy and round window membrane insertion or cochleostomy, if we have to. In cases with very laterally placed vertical segment of the facial nerve a trans- mastoid trans- attic approach used with trans canal monitoring as an alternative approach. Position of the vertical segment of the facial nerve (VFN) determined by coronal view HRCT of temporal bone, bone window of 0.6 mm thickness by using the cut posterior to the internal auditory canal at the level of lateral semicircular canal (LSCC) and then drawing a line parallel to the bony canal of the VFN and another parallel line on the outer bony wall of lateral semicircular canal (LSCC), and comparing level of both. The location of the facial nerve classified into normal if the FN is medial, same level or lateral to LSCC . Investigators referred the laterally placed FN (LPFN) when the whole vertical segment of facial nerve is lateral to LSCC. In addition, distance between VFN and LSCC was measured in cases of laterally placed FN.

Investigators proposed a radiological classification system of the mastoid segment of facial nerve to predict round window niche accessibility through posterior tympanotomy pre-operatively by using coronal view computed tomography scan of temporal bone. Facial nerve position classified into 3 types in relation to LSCC:

1. TYPE I Medial to LSCC
2. TYPE II Same level of LSCC
3. TYPE III Laterally placed to LSCC III a) Less than 2mm III b) More than 2mm

ELIGIBILITY:
Inclusion Criteria:

* All patient who underwent cochlear implant surgery with preoperative computed tomography scan and high resolution CT scan of temporal bone

Exclusion Criteria:

* None

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients admitted to otorhinolaryngology department at king Fahad Hospital of University
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2010-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Radiological classification of vertical segment of facial nerve | 48 hours before surgery
  - Radiological classification of vertical segment of facial nerve by studying temporal bone CT scan using an implemented scoring system
  1. TYPE I Medial to LSCC
  2. TYPE II Same level of LSCC
  3. TYPE III Laterally placed to LSCC III a) Less than 2mm III b) More than 2mm

SECONDARY OUTCOMES:
Surgical approach in cochlear implantation | For 4 hours after start of surgery
  The surgical approach used for cochlear implantation

CONTACTS AND LOCATIONS:
Overall Officials: Laila M Al Telmesani, MD, Principal Investigator — ENTDepartment, Dammam University, Dammam, Saudi Arabia
Locations (1):
- Dammam University KFHU, Khobar, EP, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided